CLINICAL TRIAL: NCT05612711
Title: Single-site, Randomized, Double-Blind, Placebo-Controlled Crossover Trial of Dronabinol for the Treatment of Agitation in Outpatient With Dementia
Brief Title: Dronabinol for Agitation in Dementia Crossover Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not funded
Sponsor: Ralph H. Johnson VA Medical Center (U.S. Federal Agency)
Collaborators: JHSPH Center for Clinical Trials (Other)
Responsible Party: Principal Investigator, Jacobo Mintzer, MD, Professor, Geriatric Psychaitrist, Ralph H. Johnson VA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1I01CX002671
Record Dates: First submitted 2022-10-28; First posted 2022-11-10 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Dementia Moderate; Dementia Severe; Agitation,Psychomotor; Behavioral Symptoms
Keywords: Dementia; Agitation; Behavioral and Psychological Symptoms of Dementia
MeSH Terms: conditions — Psychomotor Agitation; Behavioral Symptoms; Dementia; Behavior | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomization to either dronabinol or placebo (1:1 assignment ratio) for a total of 8 weeks (1 week of titration, followed by 6 weeks of treatment at target dose, followed by 1 week of taper). All subjects will then undergo a 3-week placebo washout phase, followed by the crossover intervention for 8 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug vs placebo filler will be "over-encapsulated" for masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dronabinol First (Experimental): Participants will take Dronabinol 2.5 mg capsules twice daily for 1 week, followed by dronabinol 5 mg twice daily for 6 weeks, followed by dronabinol 2.5 mg twice daily for 1 week. They will then undergo a 3-week washout period, followed by placebo capsules twice daily for 8 weeks.
  Interventions: Drug: Dronabinol
- Placebo First (Experimental): Participants will take matching placebo capsules twice daily for 8 weeks, followed by a three week washout period. They will then begin taking dronabinol 2.5 mg capsules twice daily for 1 week, followed by dronabinol 5 mg twice daily for 6 weeks, followed by dronabinol 2.5 mg twice daily for 1 week.
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — All participants will take both dronabinol and placebo at different points in the study in this crossover design trial.
  Other Names: Marinol

SUMMARY:
The goal of this clinical trial is to study the effects of dronabinol in US Veterans with agitation related to moderate to severe dementia. The main goals of the study are:

* To evaluate the efficacy of dronabinol for the treatment of agitation in moderate to severe dementia compared to placebo
* To evaluate the safety of dronabinol in the treatment of agitation in moderate to severe dementia compared to placebo

Fifty (50) subjects will be given either dronabinol or placebo for 8 weeks. All subjects will then undergo a "washout" phase for 3 weeks, followed by the crossover intervention (i.e. subjects who received placebo during the first phase will receive dronabinol during the second phase, and vice versa). Thus, all participants will be taking dronabinol at some point during the study. During the study, subjects will undergo evaluations for:

* Agitation
* Cognitive changes
* Physical changes (i.e. labs, ekg, physical exam)

DETAILED DESCRIPTION:
The investigators will conduct a phase IIa study to evaluate the efficacy and safety of dronabinol in the treatment of agitation related to dementia in the US Veteran population.

Specific Aim 1 - To evaluate the efficacy of dronabinol (target dose 5 mg bid) for the treatment of agitation in dementia.

Hypothesis: Dronabinol improves clinically significant agitation in moderate to severe dementia. Approach: The investigators will conduct a 6-week, double-blind, placebo-controlled, crossover, exploratory study of 50 Veterans suffering from moderate to severe dementia and clinically significant agitation with the Cohen Mansfield Agitation Inventory (CMAI) total score as the main outcome measure. Impact: The potential benefit of dronabinol in agitation will be evaluated.

Specific Aim 2 - To evaluate the safety of dronabinol in the treatment of agitation in moderate to severe dementia.

Hypothesis: Dronabinol is safe for the treatment of agitation in moderate to severe dementia. Approach: Outcomes of safety monitoring are to be measured by physical examination, vital signs with weight, adverse event reports, electrocardiogram, safety labs including complete metabolic panel (CMP), complete blood count (CBC), urinalysis (UA), and treatment compliance. Impact: The potential adverse effects of the 5 mg dose of dronabinol will be evaluated.

Exploratory Aims - The investigators will also evaluate the effect of dronabinol on neuropsychiatric symptoms, caregiver distress, cognition, weight, nutritional status, pain, and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* US Veteran who is not pregnant or unable to become pregnant
* Diagnosis of Major Neurocognitive Disorder (aka dementia) of any type
* Functional Assessment Staging Test (FAST) score of 5 or higher
* Presence of clinically significant agitation and/or irritability with an NPI subscale score greater than or equal to 4
* If treated with cholinesterase inhibitors or memantine, dosage must be stable for 3 months, or if discontinued they may enroll after 1 month
* Must be able to swallow capsules
* Must meet International Psychogeriatric Association's provisional definition of agitation in dementia.
* Must have decisional capacity to sign informed consent or have a legally authorized representative available to provide consent
* Must have an available study partner who spends at least 10 hours per week with the subject.

Exclusion Criteria:

* Psychotropic medication changes (i.e. concomitant antidepressants, antipsychotics) less than 1 month prior to study randomization
* Contraindications to dronabinol (hypersensitivity or allergy to any cannabinoid or sesame oil)
* Use of cannabinoids (including over the counter products such as "CBD" or medical cannabis) or other illicit drugs in the past 3 months
* History of psychotic symptoms due to another psychiatric illness other than dementia int he past 2 years.
* Unstable current psychiatric disorder or neurologic condition (i.e. unstable depression, bipolar disorder, epilepsy, etc.) other than agitation or psychosis due to dementia.
* Suicidal ideations in the past 3 months or attempts in the past year
* Clinically significant delusions and/or hallucinations which are considered by the PI's to be a contraindication for dronabinol use
* Taking 1 or more medications which in the judgement of the PI's can be contraindicated with the use of dronabinol
* Unstable or uncontrolled medical conditions including cardiovascular system issues (i.e. angina, cardiac arrhythmias, recurrent syncope, hypertension, etc) as judged by the PI's.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in agitation, Cohen Mansfield Agitation Inventory (CMAI) | Baseline (0 weeks) to 18 weeks
  A 29-item scale to assess 4 dimensions of agitation across a range of frequencies during the previous two weeks. Scores range from 29-203, where higher scores indicate greater agitation severity.
Safety and tolerability, Treatment Emergent Adverse Events | Baseline (0 weeks) to 18 weeks
  We will compare the frequency of reported adverse events using Common Terminology Criteria for Adverse Events version 4.0

SECONDARY OUTCOMES:
Change in agitation, Neuropsychiatric Inventory (NPI) | Baseline (0 weeks) to 18 weeks
  This scale provides a comprehensive evaluation of neuropsychiatric symptoms in the previous month across 12 domains of behavior. Total scores range from 0-144, where higher scores reflect a greater level of neuropsychiatric symptom burden.
Change in caregiver distress, Neuropsychiatric Inventory - Caregiver distress score | Baseline (0 weeks) to 18 weeks
  Caregiver distress is rated for each positive neuropsychiatric symptom domain on a scale of 0 (not distressing at all) to 5 (extremely distressing). Thus total scores range from 0-60 on for the 12 domains.
Clinically perceptible effect of dronabinol on agitation, modified Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (mADAS-CGIC) | Baseline (0 weeks) to 18 weeks
  This modified version of the Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change assesses ites specific to agitation in Alzheimer's disease to produce a global rating of change in agitation and a measure of clinical significance. Scores range from 1 to 7 where 1 = marked improvement, 4 = no change, and 7 = marked worsening)
Change in cognition, standardized Mini Mental Status Examination (sMMSE) | Baseline (0 weeks) to 18 weeks
  The standardized version of the original MMSE is a 30 point scale to measure global cognition, where lower scores indicate greater cognitive impairment.
Change in cognition, Alzheimer's Disease Assessment Scale - Cognitive Section (ADAS-Cog) | Baseline (0 weeks) to 18 weeks
  This scale includes 11 items, 8 of which are performance based and 3 are ratings of language impairment. Scores range from 0-70, where higher scores indicate greater impairment. This scale will be administered to subjects scoring greater than or equal to 12 on the sMMSE.
Change in cognition, Severe Impairment Battery | Baseline (0 weeks) to 18 weeks
  The severe impairment battery is a measure of cognition developed for the evaluation of patients whose dementia severity is such that they cannot complete conventional neuropsychological testing. It will be administered to anyone with an sMMSE score less than 12. Scores range from 0 to 133, where lower scores indicate greater impairment.
Change in nutritional status, prealbumin | Baseline (0 weeks) to 18 weeks
  Assessed by changes in prealbumin (mg/dl)
Change in nutritional status, weight | Baseline (0 weeks) to 18 weeks
  Assessed by changes in weight (kg)
Change in pain, Pain Assessment in Advanced AD (PAIN-AD) scale | Baseline (0 weeks) to 18 weeks
  The PAIN-AD scale is a 5-item rater observed scale to measure pain in patients with dementia. Scores range from 0-10, where higher scores suggest a higher level of pain.
Change in blood pressure | Baseline (0 weeks) to 18 weeks
  Blood pressure (mm Hg) will be monitored every 2 weeks
Change in heart rate | Baseline (0 weeks) to 18 weeks
  Heart rate will be monitored in beats per minute (bpm) every 2 weeks to monitor safety.
Change in QTc interval on Electrocardiogram (EKG) | Baseline (0 weeks) to 18 weeks
  EKGs will be monitored at each study visit to assess changes in QTc interval and monitor safety

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo E Mintzer, MD, Principal Investigator — Ralph H. Johnson VA Healthcare System; Jessica E Broadway, MD, Principal Investigator — Ralph H. Johnson VA Healthcare System
Locations (1):
- Ralph H. Johnson VA Health Care System, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No